CLINICAL TRIAL: NCT04520503
Title: Relationship Between Pre-induction Electroencephalogram Pattern of Adult Patients and Their Sensitivity to Propofol
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Professor (full), Seoul National University Hospital
Other Study IDs: pre-induction EEG
Record Dates: First submitted 2020-08-05; First posted 2020-08-20 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Propofol Overdose of Undetermined Intent
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pre EEG group: This cohort includes all participants in this study. EEG sensor will be attached to the patient's forehead before induction of anesthesia. Patterns of EEG and data will be obtained
  Interventions: Drug: Propofol; Device: EEG monitoring

INTERVENTIONS:
Drug: Propofol — The dose of propofol required for loss of consciousness and the total induction dose of propofol will be recorded for every patients.
Device: EEG monitoring — The processed EEG spectrogram and indices, such as patient status index, 95% spectral edge frequency, and suppression ratio, will be obtained from Sedline monitoring device. The raw pre-induction EEG will be extracted from Sedline at the end of induction and it will be analyzed by an external software to calculate the mean frequency, frequency band power and its distribution.

SUMMARY:
The induction dose of propofol is generally determined based on patients' characteristics, underlying disease, general condition, and also by clinician's experiences. However, It is difficult to anticipate and objectively calculate an adequate dose of propofol for every patient considering the variability of an individual's response to propofol. If there is a specific pattern in EEG prior to induction of anesthesia that can provide information about the patient's susceptibility to propofol, every induction may be performed far more smoothly with a precisely optimized dose of propofol for each patient. The study is to find a relationship between the pre-induction EEG pattern of adult patients and their sensitivity to propofol.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing general anesthesia

Exclusion Criteria:

* Patients undergoing cardiac or brain surgery
* Patients with neurological deficit or impaired communication (Glasgow Coma Scale < 15)
* Unstable vital sign (cardiogenic, hemorrhagic, septic shock)
* Patients with eclampsia
* Patients who administered preoperative anxiolytics
* Patients who do not require intubation
* Patients who are considered unsuitable for the study

Ages: 20 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients, who are aged between 20 and 89 years old, undergoing general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Absolute and Relative power in distinct frequency (% δ: 1-4 Hz, % θ: 5-8 Hz, % α: 9-12 Hz, % β: 13-25 Hz) | During the induction of anesthesia (up to 15 min)
  Relative power in distinct frequency (% δ: 1-4 Hz, % θ: 5-8 Hz, % α: 9-12 Hz, % β: 13-25 Hz)
Processed EEG index (PSI; patient state index) | During the induction of anesthesia (up to 15 min)
  Processed EEG index (PSI; patient state index)
Mean frequency and 95% spectral edge frequency (Hz) | During the induction of anesthesia (up to 15 min)
  Mean frequency and 95% spectral edge frequency (Hz)
Burst suppression ratio (%) | During the induction of anesthesia (up to 15 min)
  Burst suppression ratio (%)

SECONDARY OUTCOMES:
The effect-site concentrations of propofol at loss of consciousness (μg/ml) | During the induction of anesthesia (up to 15 min)
  The effect-site concentrations of propofol at loss of consciousness (μg/ml)
The dose of propofol required for loss of consciousness (mg) | During the induction of anesthesia (up to 15 min)
  The dose of propofol required for loss of consciousness (mg)
Total amount of propofol used (mg) | During the induction of anesthesia (up to 15 min)
  Total amount of propofol used (mg)
Time to loss of consciousness (second) | During the induction of anesthesia (up to 15 min)
  Time to loss of consciousness (second) after the start of induction
Vital sign - blood pressure | During the induction of anesthesia (up to 15 min)
  Check blood pressure (mmHg)
Vital sign - heart rate | During the induction of anesthesia (up to 15 min)
  Check heart rate (beats per minute)
Administration of vasopressors (ephedrine, phenylephrine, epinephrine, etc) | During the induction of anesthesia (up to 15 min)
  Administration of vasopressors (ephedrine (mg), phenylephrine (mcg), epinephrine (mcg), etc)

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided